CLINICAL TRIAL: NCT04309227
Title: Comparison of Traditional High-Load Training With Low-Load Plus Blood Flow Restriction Training on Strength, Function, and Self-Reported Outcomes in Patients With Rheumatoid Disorders
Brief Title: Comparison of Training Load With/Out Blood Flow Restriction Training in Rheumatoid Populations
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of participant recruitment; closure of study based on investigator feedback
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00001312
Record Dates: First submitted 2020-02-28; First posted 2020-03-16 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2023-10

CONDITIONS: Rheumatoid Arthritis; Myositis; Osteoarthritis; Weakness, Muscle
Keywords: rheumatoid arthritis; osteoarthritis; myositis; blood flow restriction; strength training; weight training
MeSH Terms: conditions — Arthritis, Rheumatoid; Myositis; Osteoarthritis; Muscle Weakness | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator responsible for outcomes assessment and evaluation will be blinded. The investigator performing statistical analysis will not be involved with any interventions or assessments prior to being provided data.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional High-Intensity Training (Experimental): Participants will perform their training at ~70% of their 1-repetition maximum, as traditionally advocated in strengthening literature. Each of the diagnoses (RA, OA, myositis) will have a High-Intensity arm.
  Interventions: Other: Strength Training
- Low Intensity plus Blood Flow Restriction Training (Experimental): Participants will perform their training at ~30% of their 1-repetition maximum, and will have blood flow partially occluded (60-70%) to the training limb. Each of the diagnoses (RA, OA, myositis) will have a Low-Intensity plus Blood Flow Restriction arm.
  Interventions: Other: Strength Training
- Control (No Intervention): Each of the diagnoses (RA, OA, myositis) will have a control arm. The control groups will be evaluated at time 0, 4 weeks, and 8 weeks but will not receive intervention.

INTERVENTIONS:
Other: Strength Training — Strength training traditionally requires use of high intensity loads to stimulate muscle growth and strength improvements. Some participants will be randomized to a traditional strength training program.
  Blood Flow Restriction (BFR) training is used to stimulate muscle hypertrophy and strength improvements in a variety of populations. Results of BFR training are comparable to traditional high intensity training (HIT) despite using weight that are at a low intensity (low percent of 1 repetition maximum). This intervention has not been extensively studies in the rheumatoid or osteoarthritis populations, nor the myositis populations despite idealogical benefit for each group of low-load strengthening.
  Arms: Low Intensity plus Blood Flow Restriction Training; Traditional High-Intensity Training

SUMMARY:
The study will investigate the effects of a traditional, high-intensity strengthening program compared to an investigational low-intensity strengthening program that also uses blood flow restriction as part of the training program. Both groups will be compared to a control group, which will receive no training. Measures of strength, function, and patient outcomes will be taken before starting the training, at mid-term, and at the end of the 8-week training program. Additionally, investigators will collect outcome data at 6 and 12 months after completing the program to assess for long term outcomes. The eligible populations are participants with rheumatoid arthritis (RA), osteoarthritis (OA), or myositis. The study will include about 15 participants per group, or 45 people with each diagnosis.

DETAILED DESCRIPTION:
This study is a randomized controlled trial to compare the effectiveness of low-intensity training with blood flow restriction (LIT+BFR) vs high-intensity training (HIT) vs a control group in people with RA, myositis, and osteoarthritis. Participants of each population will be randomized into LIT+BFR, HIT, or control. All functional testing and interventional procedures will be performed at the School of Allied Health Professions (SAHP). The evaluator will be blinded to group allocation. Blood draws and analysis will be performed during visits with the participant's rheumatologist at the Ambulatory Care Center, as part of the standard of care for their visits with their rheumatologist.

All participants will perform informed consent, which will take place at the SAHP Faculty Clinic. Once a participant has consented, he/she will participate in two familiarization sessions at least 48 hours apart. Familiarization sessions are designed to introduce patients to the exercise equipment, and will consist of the tests used in the evaluation portion of the intervention. Familiarization sessions also aide in better obtaining a patient's 1 repetition max (1RM, i.e. the maximum amount a person can lift one time) by decreasing the learning effect. It has a similar effect with the other functional or objective measures such as grip strength and pain-pressure threshold to decrease learning effect.

Once 1RM is determined (see 1RM test below), participants will be ranked in tertiles according to their 1RM in the leg press exercise and will then be randomly assigned to LIT+BFR, HIT, or control group. Randomization will be performed by Excel random generator. All participants will then undergo pre-testing that will include subjective questionnaires, and functional testing. Lab work will be performed by the rheumatologists as part of a participant's routine exam during the screening visit.

Investigators responsible for blood work and lab values will be blinded to participant allocation. A licensed and trained physical therapist, blinded to participant allocation, will be responsible for performing the functional tests. Testing will take a place on a separate day from the interventions. Due to the exercise-based intervention, participants will not be blinded to group allocation.

Prior to functional testing, each participant's blood pressure and heart rate will be measured to ensure safety with testing.

1RM test: participants will warm-up for 5 minutes on a stationary cycle. They will perform two light warm-up sets separated by a 2 minute rest. In the first set, participants will perform 8 repetitions of an estimated 50% 1RM. The second set of 8 will be adjusted to 70% 1RM. Participants will then have up to 5 attempts to achieve 1RM load with a 3 minute rest interval between attempts. 1RM test will be conducted on the leg press machine and knee extension machine.

The below outcome measures will be performed on all patient populations:

Pain: will be quantified at pre-testing and prior to each exercise session using the numeric pain rating scale. The participant will be asked to rank his/her current pain level and pain intensity in the last 24 hours.

Pain Pressure Threshold (PPT): the minimum force necessary to induce pain. PPT will be measured using a pressure algometer prior to exercise and post exercise 1 time per week at the proximal forearm and at the proximal tibialis anterior.

Rating of Perceived Exertion (RPE): Scale used to measure an individual's perceived intensity of the exercise. This will be measured after each exercise session.

Walking ability, including balance, gait speed, endurance, and fall risk will be assessed using the Timed Up and Go (TUG), 10 meter walk, and 6 minute walk test (6MWT).

Grip strength: will be measured using a handheld dynamometer. Three trials per hand will be performed and averaged with 1 minute of rest between trials.

Bicep strength: will be measured using a handheld dynamometer. Three trials per arm will be performed and averaged with 1 minute rest between trials.

Short-Form 36 (SF-36): a generic outcome survey to quantify health status and health-related quality of life. A higher score indicates better health condition with 100 being the maximum score.

Health Assessment Questionnaire (HAQ): is a patient reported outcome questionnaire and is used to measure disability in patients with rheumatoid arthritis.

The below will only be given to patients with rheumatoid arthritis:

Clinical Disease Activity Index (CDAI): is a composite score of 4 parameters: tender and swollen joints, and a patient's and physician's global score of disease activity. This will be completed by the rheumatologist before and after the study.

The below will only be given to patients with osteoarthritis:

Knee injury and osteoarthritis outcome score (KOOS): a general assessment questionnaire regarding patient's opinion on their knee pain and associated problems. To be used for participants with knee OA.

Hip Disability and Osteoarthritis Outcome Score (HOOS): a general assessment questionnaire regarding patient's opinion on their hip pain and associated problems. To be used for participants with hip OA.

Foot and Ankle Osteoarthritis Outcome Score (FAOS): a general assessment questionnaire regarding patient's opinion on their foot or ankle pain and associated problems. To be used for participants with foot or ankle OA.

Once a participant in the LIT+BFR or HIT has completed pre-testing and familiarization, he/she will return within one week to begin the exercise protocol. Participants in the control group will be advised to continue with their regular daily activity and will not return until reassessment testing at week 4 and then end of the study at week 8. Participants in LIT+BFR and HIT will come to the SAHP Faculty Clinic to perform their designated exercise program two times per week for 8 weeks. Prior to each exercise session, a participant's blood pressure and heart rate will be documented to ensure safety with proceeding with exercise. Heart rate and blood pressure will be logged and kept in a binder. Each participant's exercise program will be led by a trained research assistant or licensed physical therapist. A licensed physical therapist trained in blood flow restriction training and operation of the Delfi tourniquet system will be onsite for any questions or concerns that may arise during a participant's exercise program. Each participant will perform a standard set of exercises which is outlined below. Each participant will have the BFR cuff placed at the proximal thigh on the affected limb; only those in the LIT+BFR arm of the study will have the cuff inflated:

* Warm up: recumbent bike or stepper with or without blood flow restriction depending on allocation for 10 minutes.
* Knee extension machine (bilateral)
* Leg press (bilateral)

During the first week of training, participants will be introduced to the training load. Participants in the LIT+BFR will perform 20% of their 1RM and participants in HIT will perform 50% of 1RM. During the 2nd week of training intensity will be adjusted to 30% 1RM and 70% 1RM for LIT+BFR and HIT respectively. LIT+BFR will perform 1 set of 30 repetitions upon initiating weighted exercise (i.e. knee extension machine and leg press machine). After the completion of 30 repetitions of the respective exercise, he/she will perform an additional 3 sets of 15 repetitions. The HIT group will perform 4 sets of 10 repetitions of each respective exercise. A one minute rest will be allowed between all sets for each group

1RM will be reassessed at 4 weeks and training loads will be adjusted accordingly.

Blood flow restriction for participants in the LIT+BFR will be determined by the Delfi system. A full description of the Delfi system can be found in section 9.4. Briefly, a specialized blood pressure cuff will be applied to the proximal thigh prior to the start of each session. The Delfi system will measure the participant's full occlusion pressure and will then be adjusted to 80% of full occlusion to begin the exercise protocol. The occlusion pressure will be maintained throughout the exercise and will be relieved (reperfusion phase) after the completion of all sets of each individual exercise. The participant will be allowed to rest for up to 3 minutes between exercises. If a participant verbalizes discomfort, the occlusion pressure will be decreased and/or the repetitions or sets will be decreased. Participants will be allowed to stop the exercise protocol at any time should they experience significant discomfort.

A participant will be considered to have completed the study after participating in 8 weeks of exercise training with at least 12 of 16 intervention visits. At the end of the training protocol, the participant will again come to the SAHP Faculty Clinic within one week of study completion for post-testing. He/she will complete the questionnaires and functional testing as noted for pre-testing. He/she will go to the Rheumatology Clinic to complete routine blood work/lab values. Participants in the control group will come back for post testing after 8 weeks of continuing usual daily activity.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis from LSUHSC-SHreveport Rheumatologist of rheumatoid arthritis (RA), osteoarthritis (OA), or myositis
* stable medication for at least 3 months
* OA in weightbearing joints, and limited to non-advanced OA per Kellgren Lawrence grading
* cleared by rheumatologist for participation in high intensity training and blood flow restriction training

Exclusion Criteria:

* cardiovascular or other disease preventing exercise participation
* within past 6 months, have performed regular physical activity training or physical therapy
* one or more arthroplasty in weight-bearing joints
* taking more then 5mg of prednisone in past 3 months
* unable to perform timed up and go test, 10 meter walk test, or 6 minute walk test without more than supervision assistance; assistive devices can be used

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
lower extremity strength | Lower extremity strength tests are performed at 0, 4, and 8 weeks, and should take 15-20 minutes to complete
  Participant's leg strength will be measured by performing a one-repetition maximum lift on both the leg press and leg extension machines. This will be measured at the start of the study, and reassessed with a percent change determined at 4 and 8 weeks. The leg strength measurements will be used to set the weight used during exercise interventions.
Functional Strength by the Timed-up-and-Go test | The Timed-up-and-Go will be performed at 0, 4, and 8 weeks and should take 2 minutes to complete.
  Participants will perform the Timed-up-and-Go test, which consists of standing up from a chair, walking a short distance, turning, and returning to the chair. Participants are timed on how long this task takes, and it has been validated as a measure of functional leg strength and balance. The test will be performed when starting the study, and reassessed at 4 and 8 weeks.
Gait Speed | Gait speed is performed at 0, 4, and 8 weeks and should take 2 minutes to complete.
  Participants will be timed on how quickly they are able to walk 10 meters, which will be used to calculate their gait speed in meters per second. The test will be performed when starting the study, and reassessed at 4 and 8 weeks.
Health Assessment Questionnaire | The HAQ is performed at 0, 4, and 8 weeks; repeated 6 and 12 months post-intervention, and should take 10-20 minutes to complete.
  The Health Assessment Questionnaire (HAQ) asks a series of questions regarding how participants view their health. Each question is rated from 0-3, with a higher score indicating higher levels of disability. The HAQ is used in this study to investigate changes in self-perceived health status. It will be given on initial visit, and repeated at 4 and 8 weeks. It will be given again as part of the long-term follow-up at 6 and 12 months post-intervention.
Cardiovascular endurance walking test | The 6 minute walk test is performed at 0, 4, and 8 weeks, and should take 6 minutes to complete.
  Participants will perform the 6-minute walk test as a measure of cardiovascular endurance. The test involves walking a track for 6 minutes, with instructions to walk as fast as possible for the whole 6 minutes. Distance walked will be recorded and compared to normal values. The test will be performed when starting the study, and reassessed at 4 and 8 weeks.

SECONDARY OUTCOMES:
Self-Reported function | Short Form-36 is completed at 0, 4, and 8 weeks; repeated 6 and 12 months post-intervention. It should take 10-20 minutes to complete.
  Short Form-36 questionnaire will also be used to measure overall self-reported function. The Short Form-36 questionnaire has 8 sub-scales examining different aspects of function, with each sub-scale scored 0-100. A higher score indicates better function.
Self-Reported function in patients with hip osteoarthritis (OA) | The HOOS is completed at 0, 4, and 8 weeks; repeated 6 and 12 months post-intervention. It should take 10-20 minutes to complete.
  The Hip Osteoarthritis Outcome Score (HOOS) examines self-reported function related to osteoarthritis symptoms in the hip. It is scored from 0-100, with a higher score indicating better function. The test will be performed when starting the study, and reassessed at 4 and 8 weeks, and then at long-term follow up at 6 and 12 months post-intervention. A change score will be calculated with each reassessment.
Self-Reported function in patients with knee osteoarthritis (OA) | The KOOS is completed at 0, 4, and 8 weeks; repeated 6 and 12 months post-intervention. It should take 10-20 minutes to complete.
  The Knee Osteoarthritis Outcome Score (KOOS) examines self-reported function related to osteoarthritis symptoms in the knee. It is scored from 0-100, with a higher score indicating better function. The test will be performed when starting the study, and reassessed at 4 and 8 weeks, and then at long-term follow up at 6 and 12 months post-intervention. A change score will be calculated with each re-assessment.
Self-Reported function in patients with foot and/or ankle osteoarthritis (OA) | The Foot and Ankle Outcome Score is completed at 0, 4, and 8 weeks; repeated 6 and 12 months post-intervention. The Foot and Ankle Outcome Score
  The Foot and Ankle Outcome Score examines self-reported function related to osteoarthritis symptoms in the foot and/or ankle. It is scored from 0-100, with a higher score indicating better function. The test will be performed when starting the study, and reassessed at 4 and 8 weeks, and then at long-term follow up at 6 and 12 months post-intervention. A change score will be calculated with each re-assessment.
Clinical Disease Activity Index (CDAI) | This assessment will be performed by the physician pre/post intervention, and should take 10 minutes to complete.
  The CDAI is completed by the rheumatologist for participants with rheumatoid arthritis only. It will assess the number of tender and swollen joints, the patient's global score of disease activity, and the physician's global assessment of disease activity. One composite score is calculated, with a high score of 76 indicating high disease activity and a low score of 0 indicating remission.
Biceps muscle strength | Biceps strength tests are performed at 0, 4, and 8 weeks and should take 2 minutes to complete
  Biceps strength will be measured using a hand-held dynamometer, which measures how much force the participant is able to resist using their biceps muscle. Biceps strength will be tested when the participant initially starts the study, and then reassessed at 4 and 8 weeks. At each reassessment, a percent change in biceps strength will be calculated.
Grip Strength | Grip strength measurements are performed at 0, 4, and 8 weeks, and should take 2 minutes to complete
  Grip strength will be measured using a dynamometer that measures how strong the participant is able to squeeze the dynamometer. Biceps strength will be tested when the participant initially starts the study, and then reassessed at 4 and 8 weeks. At each reassessment, a percent change in biceps strength will be calculated.
Numeric Pain Rating Scale | numeric pain rating scale will be rated at every participant encounter, and takes less than 1 minute to complete.
  Pain will be assessed using the numeric pain rating scale. Scores range from 0-10, with higher scores indicating higher levels of pain.
Pain Pressure Threshold | Pain pressure threshold will be measured one time per week, and is estimated to take 2 minutes to complete.
  The Pain Pressure Threshold is measured by gradually applying more pressure to an area of the skin using a pressure algometer. The participant is instructed to report when the sensation changes from pressure to pain. The pounds of pressure applied is measured with the algometer and recorded. This measurement will be assessed at the upper extremity along the distal forearm, and lower extremity at the proximal anterior tibialis muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Erin McCallister, DPT, Principal Investigator — LSUHSC-Shreveport
Locations (1):
- LSUHSC-Shreveport, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Will not be shared outside of investigators

REFERENCES:
- [Background] Rodrigues R, Ferraz RB, Kurimori CO, Guedes LK, Lima FR, de Sa-Pinto AL, Gualano B, Roschel H. Low-Load Resistance Training With Blood-Flow Restriction in Relation to Muscle Function, Mass, and Functionality in Women With Rheumatoid Arthritis. Arthritis Care Res (Hoboken). 2020 Jun;72(6):787-797. doi: 10.1002/acr.23911. Epub 2020 May 14. PMID 31033228
- [Background] Mattar MA, Gualano B, Perandini LA, Shinjo SK, Lima FR, Sa-Pinto AL, Roschel H. Safety and possible effects of low-intensity resistance training associated with partial blood flow restriction in polymyositis and dermatomyositis. Arthritis Res Ther. 2014 Oct 25;16(5):473. doi: 10.1186/s13075-014-0473-5. PMID 25344395
- [Background] Santos AR, Neves MT Jr, Gualano B, Laurentino GC, Lancha AH Jr, Ugrinowitsch C, Lima FR, Aoki MS. Blood flow restricted resistance training attenuates myostatin gene expression in a patient with inclusion body myositis. Biol Sport. 2014 Jun;31(2):121-4. doi: 10.5604/20831862.1097479. Epub 2014 Apr 5. PMID 24899776
- [Background] Gundermann DM, Walker DK, Reidy PT, Borack MS, Dickinson JM, Volpi E, Rasmussen BB. Activation of mTORC1 signaling and protein synthesis in human muscle following blood flow restriction exercise is inhibited by rapamycin. Am J Physiol Endocrinol Metab. 2014 May 15;306(10):E1198-204. doi: 10.1152/ajpendo.00600.2013. Epub 2014 Apr 1. PMID 24691032
- [Background] Karabulut M, Sherk VD, Bemben DA, Bemben MG. Inflammation marker, damage marker and anabolic hormone responses to resistance training with vascular restriction in older males. Clin Physiol Funct Imaging. 2013 Sep;33(5):393-9. doi: 10.1111/cpf.12044. Epub 2013 Apr 23. PMID 23701309
- [Background] Takarada Y, Takazawa H, Sato Y, Takebayashi S, Tanaka Y, Ishii N. Effects of resistance exercise combined with moderate vascular occlusion on muscular function in humans. J Appl Physiol (1985). 2000 Jun;88(6):2097-106. doi: 10.1152/jappl.2000.88.6.2097. PMID 10846023
- [Background] Roschel H, Neves-Junior M, Gualano B, Barroso R, Robles C, de Sa Pinto AL, Fuller R, Lima FR. Familiarisation with lower limb strength testing in middle-aged women with osteoarthritis of the knee. Physiotherapy. 2011 Dec;97(4):350-3. doi: 10.1016/j.physio.2011.01.007. Epub 2011 Apr 15. No abstract available. PMID 22051593
- [Background] Brown LE WJ. Accurate assessment of muscular strength and power. Journal of Exercise Physiology Online. 2001;4(1):1-21.
- [Background] Abe T HS, Beekley MD, Koizumi K. Day-to-day change in muscle strength and MRI-measured skeletal muscle size during 7 days KAATSU resistance training: A case study. Int J KAATSU Train Res. 2005;1:71-76.